CLINICAL TRIAL: NCT04613167
Title: Genetic, Biochemical and Functional Markers of Cardiovascular Risk in Patients With Premature Coronary Artery Disease and Treatment Options
Brief Title: Markers of Cardiovascular Risk in Patients With Premature Coronary Artery Disease and Treatment
Acronym: GEBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Miran Sebestjen, Professor, principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEBI
Record Dates: First submitted 2020-10-06; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Acute Coronary Syndrome; Premature Coronary Heart Disease; Lipoproteinemia; Inflammation; Genetic Polymorphisms
Keywords: Coronary heart disease; Acute coronary syndrome; Lipoprotein (a); Genetics; Secondary prevention; Endothelium; Inflammation; Genetic polymorphisms; NO synthetase; Dyslipidemia
MeSH Terms: conditions — Acute Coronary Syndrome; Inflammation; Coronary Disease; Dyslipidemias | interventions — alirocumab; evolocumab; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alirocumab (Experimental): The first group of patients will receive 150 mg of alirocumab every two weeks subcutaneously for 6 months
  Interventions: Drug: Alirocumab
- Evolocumab (Experimental): the second group of patients will receive evolocumab 140 mg every two weeks subcutaneously for 6 months
  Interventions: Drug: Evolocumab
- Control group (Experimental): Control group will be included in the treatment after 6 months. During this time, the control group will not receive treatment with alirocumab or evolocumab, only standard guidelines-based treatment
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Alirocumab — The first group will receive alirocumab. Blood samples from all patients will be drawn for laboratory measurements and genetics determination. Ultrasound measurement of endothelium-dependent dilatation of the brachial artery, intima media thickness of carotid arteries and pulse wave will be measured.
  Arms: Alirocumab
Drug: Evolocumab — The second group will receive evolocumab. Blood samples from all patients will be drawn for laboratory measurements and genetics determination. Ultrasound measurement of endothelium-dependent dilatation of the brachial artery, intima media thickness of carotid arteries and pulse wave will be measured.
  Arms: Evolocumab
Drug: Control group — The third group will receive only optimal guidelines-based secondary preventive treatment. Blood samples from all patients will be drawn for laboratory measurements and genetics determination. Ultrasound measurement of endothelium-dependent dilatation of the brachial artery, intima media thickness of carotid arteries and pulse wave will be measured.
  Arms: Control group

SUMMARY:
The aim of study is to examine the relationship between lipid subfractions, inflammation and structural-functional properties of the arterial wall in patients with premature coronary heart disease, to study genetic polymorphisms that determine lipid subfractions concentration on the functional and morphological properties of the arterial vascular wall in patients with early coronary heart disease, to study the effect of alirocumab and evolocumab on lipid subfractions, inflammation and structural-functional properties of arterial wall in patients with early coronary atherosclerosis and to study the influence of NOS-3 gene expression on the functional and morphological properties of the arterial vascular wall in the same patients. Impaired blood fat metabolism and chronic inflammation are intertwined as possible causes of atherosclerosis. Lipoprotein (a) (Lp (a)) is an important risk factor for coronary heart disease and a prognostic predictor in patients after myocardial infarction, but recent research suggests that subtilisin-kexin convertase type 9 (PCSK9) inhibitors are the only drugs that significantly reduce serum Lp (a) concentration. However, there are no data on the relationship between Lp (a) values and polymorphisms for Lp (a), indicators of inflammation and impaired arterial function, and response to treatment with various PCSK9 inhibitors in patients with early coronary heart disease.

DETAILED DESCRIPTION:
Impaired blood fat metabolism and chronic inflammation are intertwined as possible causes of atherosclerosis. Lipoprotein (a) (Lp (a)) is a specific subfraction of lipoprotein that is an independent risk factor for coronary heart disease and at the same time predicted residual risk in patients with pre-existing atherosclerosis, regardless of serum LDL-cholesterol concentration. Circulating levels of Lp(a) are mainly genetically determined and varies according to ethnic group. Lp(a) has many functions, which include atherosclerotic, prothrombotic and pro-inflammatory roles. The gene encoding apo (a); LPA, is located on the long arm of chromosome 6 (6q2,6-2,7) and most variants in Lp (a) can be explained by genetic diversity in LPA. To date, the most studied genetic variant is the Kringle-IV type-2 (KIV2) polymorphism, which explains 30-70% of the diversity in Lp (a) in the population. Some KIV2 replicates are associated with smaller isoforms and higher plasma concentrations of Lp (a) which are causally and independently associated with coronary heart disease. Within LPA, the number of KIV2 copies, as well as one nucleotide polymorphism (SNP), rs3798220 and rs10455872, is associated with Lp (a) concentration and coronary heart disease. Recently 'Proprotein convertase subtilisin/kexin type 9' (PCSK9) inhibitors that act through non-specific reduction of Lp(a) are the only drugs that have shown effectiveness in clinical trials, to provide reductions in cardiovascular morbidity and mortality. The effects of PCSK9 inhibitors are not purely through Lp(a) reduction, but also through LDL cholesterol reduction.

The early stage of the atherosclerosis process is characterized by endothelial cell damage, which results in impaired release and function of nitric oxide (NO) from the endothelium. NO is formed by endothelial NO synthetase (NOS-3) from the amino acid L-arginine, which is most pronounced in the vascular wall and is also most important in the process of atherosclerosis. The NOS-3 gene is located on chromosome 7; in the region 7q35-7q36. Functional polymorphisms are those that alter the expression or activity of NOS-3. Among them, rs2070744, rs3918226 and rs1799983 single nucleotide polymorphisms (SNP) are important. Variations in the expression and activity of NOS-3 genetic polymorphisms at exon 7 of the NOS-3 gene are associated with the incidence of myocardial infarction in very young patients who otherwise have a low atheromatous coronary artery load. Variations in the NOS-3 genes cause diversity in NO bioavailability and are responsible for endothelial dysfunction.

A 6-month observational, prospective, and randomized study will include 70 patients with a first acute coronary syndrome (ACS) (including acute transmural myocardial infarction, nontransmural myocardial infarction or unstable angina pectoris) event before age 55 and Lp (a) levels above 1000 mg / L or Lp (a) above 600 mg / L and LDL above 2.6 mmol / L. With the gradual inclusion ("step-wedge") and randomization of patients, the investigators will also provide a control group that will include 30 patients. The investigators will do anamnesis, targeted clinical examination, take blood samples for laboratory measurements, ultrasound measure endothelium-dependent dilatation of the brachial artery and intima media thickness of carotid arteries, measure pulse wave and calculate carotid artery wall stiffness. Patients will be divided into three groups according to a randomization list. The first group will receive alirocumab, the second group evolocumab, and the third group will be the control group and will be included in the treatment after 6 months. During this time, the control group will not receive treatment with alirocumab or evolocumab, only standard treatment. After 6 months, the investigators will repeat all the mentioned investigations. Patients will be informed about the purpose and course of the study before starting it. All will participate voluntarily, without pressure or inappropriate instigation, which they will confirm by signing.

The investigators hypotheses that in patients with early coronary artery disease Lp (a) and Lp (a) polymorphisms are associated with indicators of inflammation and structural-functional properties of the arterial wall; in patients with early coronary artery disease, PCSK9 inhibitors reduce the value of Lp (a), indicators of inflammation and structural and functional involvement of the arterial wall; in patients with early coronary artery disease, the influence of PCSK9 inhibitors on Lp (a), indicators of inflammation and structural-functional properties of the arterial wall depends on the presence of specific polymorphisms for Lp (a).

ELIGIBILITY:
Inclusion Criteria:

* at least 6 months after acute coronary syndrome,
* up to 55 years at the time of first acute coronary syndrome
* concentration Lp (a) above 1000 mg / L or Lp (a) above 600 mg / L and LDL above 2.6 mmol / L
* optimally treated risk factors for cardiovascular events according to currently valid guidelines.

Exclusion Criteria:

* Age <18 years or > 65 years,
* documented history of myocardial infarction less than 6 months before enrollment
* secondary dyslipidemia,
* severe renal disease (oGFR <30 ml / min),
* moderate to severe liver disease (elevated transaminases above 3 times the norm, elevated bilirubin above 2 times the norm, elevated creatinine kinase above 3 times the norm),
* acute illness 6 weeks before inclusion in the study,
* history of allergic reaction to any ingredient in the drug,
* pregnancy and lactation,
* life expectancy less than 12 months,
* unwillingness to participate or lack of availability for follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-11-10 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasound functional and morphological properties of the arterial wall and Lp (a) concentration | Baseline
  Functional and morphological characteristics of arterial wall will correlate to Lp (a) concentrations.
Concentration of Lp (a) and SNP in the LPA gene | Baseline
  The serum concentration of Lp (a) will correlate with single nucleotide polymorphisms (SNP) in the LPA gene
The effect of alirocumab or evolocumab on functional and morphological properties of arterial wall after 6 months | 6 months
  Both drugs will improve functional and morphological properties of arterial wall in with no difference between the drugs. We expect the improvements in each drug group will be in correlation with the decrease of Lp (a) concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Miran Šebeštjen, prof., Study Chair — University Medical Centre Ljubljana (Slovenia); Andreja Rehberger Likozar, MD, Principal Investigator — University Medical Centre Ljubljana (Slovenia)
Locations (1):
- University Medical Centre Ljubljana-Department of Vascular diseases and dept. of Cardiology, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rawther T, Tabet F. Biology, pathophysiology and current therapies that affect lipoprotein (a) levels. J Mol Cell Cardiol. 2019 Jun;131:1-11. doi: 10.1016/j.yjmcc.2019.04.005. Epub 2019 Apr 12. PMID 30986377
- [Background] BERG K. A NEW SERUM TYPE SYSTEM IN MAN--THE LP SYSTEM. Acta Pathol Microbiol Scand. 1963;59:369-82. doi: 10.1111/j.1699-0463.1963.tb01808.x. No abstract available. PMID 14064818
- [Background] Emerging Risk Factors Collaboration; Erqou S, Kaptoge S, Perry PL, Di Angelantonio E, Thompson A, White IR, Marcovina SM, Collins R, Thompson SG, Danesh J. Lipoprotein(a) concentration and the risk of coronary heart disease, stroke, and nonvascular mortality. JAMA. 2009 Jul 22;302(4):412-23. doi: 10.1001/jama.2009.1063. PMID 19622820
- [Background] Julius U, Tselmin S, Schatz U, Fischer S, Bornstein SR. Lipoprotein(a) and proprotein convertase subtilisin/kexin type 9 inhibitors. Clin Res Cardiol Suppl. 2019 Apr;14(Suppl 1):45-50. doi: 10.1007/s11789-019-00099-z. PMID 30838555
- [Background] Maranhao RC, Carvalho PO, Strunz CC, Pileggi F. Lipoprotein (a): structure, pathophysiology and clinical implications. Arq Bras Cardiol. 2014 Jul;103(1):76-84. doi: 10.5935/abc.20140101. PMID 25120086
- [Background] Ma L, Chan DC, Ooi EMM, Barrett PHR, Watts GF. Fractional turnover of apolipoprotein(a) and apolipoprotein B-100 within plasma lipoprotein(a) particles in statin-treated patients with elevated and normal Lp(a) concentration. Metabolism. 2019 Jul;96:8-11. doi: 10.1016/j.metabol.2019.04.010. Epub 2019 Apr 14. PMID 30995439
- [Background] Marcovina SM, Albers JJ. Lipoprotein (a) measurements for clinical application. J Lipid Res. 2016 Apr;57(4):526-37. doi: 10.1194/jlr.R061648. Epub 2015 Dec 4. PMID 26637278
- [Background] Tsimikas S. A Test in Context: Lipoprotein(a): Diagnosis, Prognosis, Controversies, and Emerging Therapies. J Am Coll Cardiol. 2017 Feb 14;69(6):692-711. doi: 10.1016/j.jacc.2016.11.042. PMID 28183512
- [Background] Clarke R, Peden JF, Hopewell JC, Kyriakou T, Goel A, Heath SC, Parish S, Barlera S, Franzosi MG, Rust S, Bennett D, Silveira A, Malarstig A, Green FR, Lathrop M, Gigante B, Leander K, de Faire U, Seedorf U, Hamsten A, Collins R, Watkins H, Farrall M; PROCARDIS Consortium. Genetic variants associated with Lp(a) lipoprotein level and coronary disease. N Engl J Med. 2009 Dec 24;361(26):2518-28. doi: 10.1056/NEJMoa0902604. PMID 20032323
- [Background] Chasman DI, Shiffman D, Zee RY, Louie JZ, Luke MM, Rowland CM, Catanese JJ, Buring JE, Devlin JJ, Ridker PM. Polymorphism in the apolipoprotein(a) gene, plasma lipoprotein(a), cardiovascular disease, and low-dose aspirin therapy. Atherosclerosis. 2009 Apr;203(2):371-6. doi: 10.1016/j.atherosclerosis.2008.07.019. Epub 2008 Jul 26. PMID 18775538
- [Background] Ober C, Nord AS, Thompson EE, Pan L, Tan Z, Cusanovich D, Sun Y, Nicolae R, Edelstein C, Schneider DH, Billstrand C, Pfaffinger D, Phillips N, Anderson RL, Philips B, Rajagopalan R, Hatsukami TS, Rieder MJ, Heagerty PJ, Nickerson DA, Abney M, Marcovina S, Jarvik GP, Scanu AM, Nicolae DL. Genome-wide association study of plasma lipoprotein(a) levels identifies multiple genes on chromosome 6q. J Lipid Res. 2009 May;50(5):798-806. doi: 10.1194/jlr.M800515-JLR200. Epub 2009 Jan 5. PMID 19124843
- [Background] Tada H, Takamura M, Kawashiri MA. Lipoprotein(a) as an Old and New Causal Risk Factor of Atherosclerotic Cardiovascular Disease. J Atheroscler Thromb. 2019 Jul 1;26(7):583-591. doi: 10.5551/jat.RV17034. Epub 2019 Apr 30. PMID 31061262
- [Background] Machado-Silva W, Alfinito-Kreis R, Carvalho LS, Quinaglia-E-Silva JC, Almeida OL, Brito CJ, Ferreira AP, Cordova C, Sposito AC, Nobrega OT; Brasilia Heart Study Group. Endothelial nitric oxide synthase genotypes modulate peripheral vasodilatory properties after myocardial infarction. Gene. 2015 Sep 1;568(2):165-9. doi: 10.1016/j.gene.2015.05.042. Epub 2015 May 20. PMID 26002446
- [Background] Hingorani AD, Liang CF, Fatibene J, Lyon A, Monteith S, Parsons A, Haydock S, Hopper RV, Stephens NG, O'Shaughnessy KM, Brown MJ. A common variant of the endothelial nitric oxide synthase (Glu298-->Asp) is a major risk factor for coronary artery disease in the UK. Circulation. 1999 Oct 5;100(14):1515-20. doi: 10.1161/01.cir.100.14.1515. PMID 10510054
- [Background] Zigra AM, Rallidis LS, Anastasiou G, Merkouri E, Gialeraki A. eNOS gene variants and the risk of premature myocardial infarction. Dis Markers. 2013;34(6):431-6. doi: 10.3233/DMA-130987. PMID 23594558
- [Background] Oliveira-Paula GH, Lacchini R, Tanus-Santos JE. Endothelial nitric oxide synthase: From biochemistry and gene structure to clinical implications of NOS3 polymorphisms. Gene. 2016 Jan 10;575(2 Pt 3):584-99. doi: 10.1016/j.gene.2015.09.061. Epub 2015 Sep 28. PMID 26428312
- [Background] Rehberger Likozar A, Zavrtanik M, Sebestjen M. Lipoprotein(a) in atherosclerosis: from pathophysiology to clinical relevance and treatment options. Ann Med. 2020 Aug;52(5):162-177. doi: 10.1080/07853890.2020.1775287. Epub 2020 Jun 8. PMID 32453609
- [Derived] Rehberger Likozar A, Levstek T, Karun T, Trebusak Podkrajsek K, Zupan J, Sebestjen M. Treatment with PCSK9 inhibitors influences microRNAs expression and changes of arterial wall properties: a randomized controlled trial. Eur J Med Res. 2025 Feb 25;30(1):138. doi: 10.1186/s40001-025-02398-6. PMID 40001082
- [Derived] Rehberger Likozar A, Ugovsek S, Sebestjen M. Effects of proprotein convertase subtilisin-kexin type 9 inhibitors on inflammatory and hemostatic parameters in post myocardial infarction patients. Eur J Pharmacol. 2024 Jan 15;963:176232. doi: 10.1016/j.ejphar.2023.176232. Epub 2023 Dec 7. PMID 38070635
- [Derived] Likozar AR, Sebestjen M. Predictors of functional and morphological arterial wall properties in coronary artery disease patients with increased lipoprotein (a) levels before and after treatment with proprotein convertase subtilisin-kexin type 9 inhibitors. Cardiovasc Ultrasound. 2023 Aug 14;21(1):15. doi: 10.1186/s12947-023-00313-9. PMID 37580777